CLINICAL TRIAL: NCT05241041
Title: Effects of Positive Psychological Group Psychotherapy and Auricular Acupressure on Gambling Severity, Withdrawal Symptoms, and Dopamine
Brief Title: Effects of Positive Psychological Group Psychotherapy and Auricular Acupressure on Withdrawal Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Inha University Hospital (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, EUN JIN LEE, Professor, Inha University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-06-012-002
Record Dates: First submitted 2021-12-14; First posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Gambling
Keywords: group counseling; acupressure; serotonin; depressive symptoms; resilience
MeSH Terms: conditions — Gambling; Depression

STUDY DESIGN:
Who Masked: Participant
Masking Description: In the first year, there is no masking to participant and researcher.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- [1st year]Auricular Acupressure Experimental Group 1 (Experimental): auricular acupressure
  Interventions: Device: auricular acupressure
- [1st year]Control Group 1 (No Intervention): education material
- [1st year]Normal Group (No Intervention): Non-gamblers
- [2nd&3rd year]Auricular Acupressure Experimental Group 2 (Experimental): auricular acupressure + group counseling
  Interventions: Behavioral: group counseling; Device: auricular acupressure
- [2nd&3rd year]Placebo Group (Placebo Comparator): placebo acupressure + group counseling
  Interventions: Behavioral: group counseling; Device: placebo acupressure
- [2nd&3rd year]Control Group 2 (No Intervention): education material

INTERVENTIONS:
Behavioral: group counseling — Group counseling with positive psychology and motivational interviewing was undertaken once per week for 6 weeks.
  Arms: [2nd&3rd year]Auricular Acupressure Experimental Group 2; [2nd&3rd year]Placebo Group
Device: auricular acupressure — Auricular acupressure using acupellets was performed for 6 weeks continuously.
  Arms: [1st year]Auricular Acupressure Experimental Group 1; [2nd&3rd year]Auricular Acupressure Experimental Group 2
Device: placebo acupressure — Placebo acupellets were prepared without metal projections, and placed on both sides in the same areas of the ear as the active condition.
  Arms: [2nd&3rd year]Placebo Group

SUMMARY:
Objective The purpose of this study is to examine the effects of auricular acupressure and group counseling with positive psychology on gambling severity, withdrawal symptoms, and dopamine.

Methods This study is a randomized controlled trial and has been performed at a University in South Korea. 180 gamblers and 60 non-gamblers will be recruited. In the first year, gamblers will be randomly assigned to two groups: Experimental Group 1 (auricular acupressure); and Control Group 1 (education material to stop and cope withdrawal symptoms). And Normal Group will be recruited independently. Furthermore, a single blind randomized controlled trial will be performed in second and third year. And gamblers will be randomly assigned to three groups: Experimental Group 2 (auricular acupressure + group counseling); Placebo Group (placebo acupressure + group counseling); and Control Group 2 (education material to stop and cope withdrawal symptoms). Auricular acupressure using acupellets is performed for 6 weeks continuously.

DETAILED DESCRIPTION:
1. Introduction The prevalence of gambling addiction is 4% in the U.S., 5.1% in South Korea. Furthermore gambling addiction causes more than 25 trillion in economic deficit annually, suicide and depression, and harmful social effects such as crime and divorce. According to a survey of 105 gambling addicts, 32.4% had depression, which is extremely high compared to 6.7% of the average person's prevalence of depression. Moreovermore, studies show that gambling addicts with depression have a higher level of addiction, childhood trauma experience, and higher nervousness and lower extroversion than those who are without depression. Gambling addicts scored higher than non-gambling addicts in anger. There is a high possibility of combined addiction and 83 studies of 11 addictions showed that gamblers were also addicted to alcohol and drugs about 36-59 percent. Those who had both gambling addiction and alcoholism had lower scores of stubbornness and cooperation compared to those who had only alcoholism. Both groups were anxious and fearful, and tended to pursue new stimuli, with low scores in self-directed areas. Online gambling addicts pursued new stimuli and showed stubborn personality traits compared to non-online gaming addicts.

   Positive psychological mediation is a way to enhance strengths or positive emotions of gratitude, honesty, love, forgiveness, resistance, faith and so on, rather than focusing on the pathological part of the subject. According to an analysis of 22 Korean studies by Nami Kim, positive psychological mediation promoted physical, subjective, psychological and social welfare, and reduced depression, anxiety symptoms, and addiction. Gratitude scores were reported to have a negative correlation with the severity of gambling. The group that wrote five grateful things for two weeks everyday increased positive sentiment, subjective happiness, and decreased negative sentiment and depression compared to the group that recorded negative things or daily life. Forgiveness reduced stresses on self-criticism, resentment and reflection on past mistakes in subjects with drug addiction and suicidal idea. The seven sessions, consisting of forgiveness, gratitude, and recall of life, reduced anxiety and depression. Psychological resilience plays a role in buffering the correlation between gambling addiction and anxiety. Positive psychological intervention has been used to treat alcoholism, internet game addiction, drug addiction, and nicotine addiction, but has never been used to treat gambling addiction.

   Auricular acupuncture is an alternative therapy that stimulates ears using seeds, magnets, stones, and metals. Furthermore, it has been used to treat nicotine and drug addiction, however, research into the problem of gambling has yet to be tried. Gambling subjects who received five weeks of body acupuncture, auricular acupuncture, auricular acupressure and counseling twice a week decreased in thrill-seeking(p=.01), gambling behaviors, ideas and desires, however, there were no statistically significant differences compared to a group who received counseling only (p=.08; effect size=0.64). As a result of applying auricular acupressure and positive psychological group counseling for quitting smoking for six weeks, withdrawal symptoms of experimental groups showed significant decrease compared to a placebo group. After a year, the smoking rate was 22.2 percent in an experimental group, 5.3 percent in a placebo group, and 5.6 percent in a control group.

   And also gamblers experience withdrawal symptoms when gamblers try to quit gamble. To begin with, a study of withdrawal symptoms in 312 gambling addicts found that 25% experienced anxiety/annoyance and 41% experienced anger, guilt and disappointment. After examining the existence of gambling withdrawal symptoms tools for this study, it is believed that it is necessary to develop them and verify reliability and validity by referring to qualitative studies on gambling withdrawal symptoms and previously developed material addiction withdrawal tools.

   Gambling addiction mechanism is as follows. Initially, gambling addiction has been reported to be linked to changes in neurotransmitters such as dopamine, serotonin and opioid. Furthermore, gamblers showed increased performance of dopamine in dynamic positron emission tomography compared to non-gambling addicts. Also, a comparison of problem and non-problem gamblers found that both groups had increased norepinephrine at the beginning of gambling, but maintained an increased norepinephrine throughout the gambling period. Meanwhile, the dopamine level of the problematic gamblers was significantly higher than that of non-problematic ones. Problematic individuals are more impulsive than those who do not have gambling problems, and blood serotonin and impulsiveness are reported to be negatively correlated.

   The auricular acupressure mechanism is as follows. Few studies have used neurotransmitters to see the effects of acupressure, and studies have shown that acupressure has altered serotonin, dopamine, epinephrine, norepine and endorphins. Subsequently, in a rat study, acupuncture for one minute a day for three days reduced alcohol withdrawal symptoms and delayed dopamine levels. Meanwhile, there are studies using self-reported questionnaires to measure the effectiveness of gambling addiction treatments, but there are only a few studies using neurotransmitters.

   The purpose of this study is to examine renouncing gambling, severity of gambling problem, withdrawal symptoms, depression, resistance, appreciation, forgiveness, serum serotonin and dopamine levels compared to those without auricular acupressure or counseling and acupressure services.
2. Method 2.1. Design and setting In the first year, the design of a study is a randomized controlled trial. And in the second and third year, the design of a study is a single blind randomized controlled trial. This study will be conducted at a University in South Korea from September 2021 to February 2025.

2.2. Sample selection Gamblers will be recruited by internet advertisement or face-to-face contacts. All gamblers will be informed about the study protocol, benefits and side effects of interventions, and the right to withdraw from the study at any time without penalty. Gamblers who agree to participate in this study will sign consent forms before data collection. Ethical approval was obtained from the institutional review board in Incheon, South Korea.

2.3. Randomization and single blinding Randomization of numbers is done by random.org to assign a number 1-60. In the first year, the researchers select the second column and a random number is generated. Following this, make a table consisting of two columns, print it out, cut out the individual numbers from the paper and put it in a nontransparent envelope and participants draw numbers from it. The ratio to be deployed to Experimental or Control Group 1 is 1:1. Normal Group is not randomly assigned. In the second and third year, the researcher will select column 3, make a table consisting of three rows, cut out the numbers from the paper, and put it in an envelope that is not visible from the outside. And participants draw numbers from it. The ratio of random assignments to experimental groups, placebo groups, and control groups is 1:1:1. There is no need for allocation of Normal Group because the participans are not recruited.

In the first year, participants will be randomly assigned to one of two groups: Experimental Group 1 (auricular acupressure); Control Group 2 (education material). Experimental and Control Group 1 know about their allocation. In the second and third year, participants will be randomly assigned to one of three groups: Experimental Group 2 (auricular acupressure + group counseling); Placebo Group (placebo acupressure + group counseling); or Control Group 2 (education material). Experimental Group 2 and Placebo Group do not know about their allocation.

2.4. Procedure The researcher will give participants website links of questionnaires to complete. Participants press a finish button to submit questionnaires after completion. All participants who apply acupellets will be instructed not to stimulate themselves with acupellets. Participants will be informed that acupellets would be changed every week, even if the acupellets fell off before the next appointment. Auricular acupressure with acupellets will be performed by the researcher mainly at Sin-moon(TF2), relaxation points (TF6), chim-jeom (LO8), head (AT2), and adrenal glands (TG2) to relieve the withdrawal symptoms on both sides, once per week for 6 weeks. Acupellets are stickers that have copper or aluminum projections. If participants will report an allergy to copper, then acupellets with aluminum projections will be applied; if participants reported an allergy to aluminum, then acupellets with copper projections were applied. If prospective participants are allergic to both copper and aluminum, then the participants will be excluded from the study.

In the second and third year, group counseling and acupressure will be performed by the researcher, who is a psychiatric-mental health nurse practitioner and an acupuncturist. Group counseling consisted of positive psychology and motivational interviewing. Each group consisted of 3-5 participants. Experimental Group 2, Placebo Group will receive group counseling for one hour per week for 6 weeks. Placebo acupellets will be prepared without metal projections, and placed on both sides in the same areas of the ear as the active condition. Auricular acupressure using acupellets will be performed for 6 weeks continuously. Group counseling and auricular acupressure will be undertaken at the same time. Control Group 2 will be encouraged not to gamble without acupressure and psychotherapy.

2.5. Data collection plan At baseline, all participants will complete general characteristics. Health history consists of onset age of gambling, current gambling frequency, amount of losses due to gambling, credit status, health problems, family history related to addiction, quitting gambling attempts, abstinence gambling intentions, and alcohol consumption. And also The Eysenck Personality Questionnaire, The Problem Gambling Severity Index (PGSI), Patient Health Questionnaire-9(PHQ-9), Adult Game Addiction Scale, Adult Smartphone Addict Diagnostic Scale, Nicotine Dependence Syndrome Scale(except Normal Group) will be completed by all participants at baseline.

Participants except Normal Group will complete The Gambling Withdrawal Scale once a week for six weeks.

PHQ-9, Korean Version of Gratitude Questionnaire, The Shortened Forgiveness Scale, Resilience, PGSI will be performed at baseline, 6 weeks, 6 months, and 1 year by Experimental Group 1 and 2, Control Group 1 and 2, and Placebo Group. Except Normal Group, Serotonin/Dopamine in the blood will be collected at baseline, 6 weeks. In Normal Group, Serotonin/Dopamine in the blood will be collected only once at baseline. And lastly, for screening Normal Group, PGSI, Adult Game Addiction Scale, Adult Smartphone Addict Diagnostic Scale, Alcohol Use Disorder Identification Test-Korea(AUDIT-K) and Urine Cotinine Test will be performed at baseline.

2.6. Sample size calculation If the investipagors put t-test, mean difference between two independent means, effect size 1, alpha 0.05, and verification power 95%, the investipagors need 54 people. A total of 60 people are needed considering the dropout rate of 10%. The effect size is 1.3, but the study is scheduled to intervene for six weeks, so the effect size is reduced to 1.

ELIGIBILITY:
[For first-year]:

Inclusion Criteria:

1. gamblers who - are more than 19 years old

   - had a total gambling period of more than six months
   * gambled within a month
   * wanted to quit gambling
   * had eight or more PGSI(Problem Gambling Severity Index) scores
   * had no ear infections
   * were not allergic to copper or aluminum
   * willing to complete questionnaires
   * agreed to extract blood
2. non-gamblers who

   * were over the age of 19
   * willing to complete questionnaires
   * agreed to extract blood
   * got zero or received the lowest scores on alcoholism, smartphone addiction, game addiction, and gambling addiction tests
   * had never smoked
   * never been blacked out in their lives
   * had negative outcome in cotinine urine tests
   * had no medical or psychological diagnosis
   * no medication for therapeutic purposes

Exclusion Criteria:

1. gamblers who - were pregnant - had experiences in taking drugs, including marijuana.
2. non-gamblers who

   * were pregnant
   * had taken painkillers in recent a week prior to blood testing
   * had experiences in taking drugs, including marijuana

[For second and third year]:

Inclusion Criteria:

1. gamblers

- will be the same as those in the first year of the study.

Exclusion Criteria:

1. gamblers who

* were undergoing gambling counseling
* were on medication
* had taken painkillers in the past a week
* were pregnant
* had experiences in taking drugs, including marijuana

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Change from Problem Gambling Severity during 1 year | baseline, 6 weeks, 6 months, 1 year
  a tool used to identify gambling addiction, with a score range of 0-27 on the Likert scale of 9 questions which require a score of 0-3. The higher the score, the more serious the gambling addiction. Scores 1-2 are classified as low risk, 3-7 as medium risk, and 8 or more as problematic gambling.
Change from Gambling Withdrawal during 1 year | baseline, 2,3,4,5,6 weeks, 6 months, 1 year
  Problem Gambling Severity Index was developed based on research into existing gambling withdrawal symptoms.The withdrawal symptoms include 14 items. Zero points have no withdrawal symptoms, one "very little" and two "nominal" and three "normal" and four "very severe". The score is between 0 and 56, and the higher the score, the worse the withdrawal symptoms. Reliability and validity will be checked in this study.
Change from serum serotonin/dopamine levels during 6 months | baseline, 6 weeks, 6 months
  A suitable sample is EDTA (WB). After calming the subjects for about 30 minutes, collect up to 12ml of peripheral blood through needles. Put the samples in an EDTA sample tube and apply them evenly on the wall of the tube, then centrifuge them for 7 minutes at 3000 rpm. Remove plasma immediately within one hour of collecting blood and store it at a temperature below minus 20 degrees Celsius.

SECONDARY OUTCOMES:
Patient Health Questionnaire-9 | baseline, 6 weeks, 6 months, 1 year
  This is a tool for measuring depression and comprises a total of nine questions. In order to find out if you have experienced depression-related problems often in the past two weeks. The score based on that zero is "none at all", one score is "three to four days", two score is "eight to ten days", three scores are "12 to 14 days", and the score is 0 to 27 and consists of a four-point scale. If the total score is more than 10 points, it is judged to have depression. In a study of 167 normal people and depressed subjects, the Chronbach's alpha coefficient was .936 and showed a high correlation with the Korean version of the Center for Epidemiological Studies Depression Scale (r=.706).
Resilience | baseline, 6 weeks, 6 months, 1 year
  This scale is an individual's inner capacity, which includes a dynamic process of heading in a more positive direction in the stress and crisis situations that an individual perceives as adversity.The 31-question tool is a four-point scale, ranging from one "not at all" to four "very much" points, with a range ranging from a minimum of 31 to a maximum of 124. The higher the score, the higher the resistance. And at the time of development, Cronbach's alpha was .85.
Korean Version of Gratitude Questionnaire | baseline, 6 weeks, 6 months, 1 year
  This tool was developed by McCullow and colleagues, and Korean Version of Gratitude Questionnaire (K - GQ - 6), which obtained reliability and validity, was measured using the Likert 7-point scale. Specifically, the scale consists of six questions: "There are so many things to be thankful for in my life," "If I list all the things I've appreciated so far," "There's not much to be thankful for in the world," "I'm grateful for many people," "I've never been more grateful for things." A single factor accounted for 56.9% of the total variations.
Korean Forgiveness Scale-Short Form | baseline, 6 weeks, 6 months, 1 year
  This form was developed by Young-hee Oh and consists of 10 questions, 4 questions that measure emotional response, 2 questions that measure cognitive response, and 4 questions that measure behavioral response. It consists of a five-point scale from 1 point "minimum" to 5 point "excessive". The range of forgiveness points is 10-50, and the higher the forgiveness score, the more forgiveness. In a study of adults, the question-to-question consistency (Cronbach's alpha) was .86, and the test-to-retest reliability for 95 college students was .78. Exploratory factor analysis and confirmatory factor analysis to determine compositional validity have shown that it is appropriate to view as one factor (explanatory variable 44.80%).
Korea Version of Alcohol Use Disorder Identification Test | baseline
  Geun-ho Cho used a tool developed by the World Health Organization (WHO) that was adapted from the Alcohol Use Disorder Identification Test(AUDIT). There are a total of 10 questions, and questions 1-8 consist of 0 to 4 points on a 5-point scale, and questions 9 and 10 score 0, 2, 4 on three scales. In Cho Geun-ho's study, the test-retest reliability was reported to be 0.93, significantly correlated with the amount of alcohol in a standard glass and the AUDIT-K score, indicating high feasibility (r=0.66 and p<0.01).
Korean Smartphone Addiction Proneness Scale for Adults | baseline
  The smartphone addiction measure was developed by National Information Society Agency in 2011. A total of 15 questions consist of four subcategories: "Daily Life Disorder", "Virtual World Experience Orientation", "Resistance", "tolerance" and "withdrawal", the score scale consists of a four-point scale from "Never" to "Excessive". The reliability Cronbach's alpha value was shown to be .81.
Korean version of Nicotine Dependence Syndrome Scale | baseline
  The nicotine-dependence syndrome scale developed by Shiffman and his colleagues (2004) was translated by Jae-woo Park(2007). As a result, it consists of 23 questions, and one point means "extremely severe" and five points means "not at all" on a five-point scale. A study of 274 health center smoking clinic participants showed confidence (internal value) of .66-90 and 8 factors in factor analysis, and 58.3% random variables described as 8 factors (Park Jae-woo, 2007).
Eysenck Personality Inventory | baseline
  This is a test that measures nine major personality dimensional factors: psychotic tendency, extroversion-introversion, adventure, impulsiveness, falseness, addiction, criminality, neurological tendency, and empathy. It consists of 121 questions, each of which is based on true and false. If the standardized T score is higher than 50, it can be interpreted as having higher scores than people of the same race and age. The Cronbach's Alpha on each scale obtained during the standardization process for Koreans was 0.65-0.87.
Urine Cotinine Test | baseline
  Cotinine urine tests will be conducted to identify non-smoking standards, which include normal groups. When smoking, nicotine is absorbed and metabolized into the body and released into urine, among which cotinine, the main metabolite, is increased in the body. The half-life of cotinine in the body is 17 hours. The manufacturer of the cotinine urine test kit to be used in the study is Hangzhou Clongene Biotech Co., Ltd., originating in China. The minimum sample amount for testing is 110microliter (3 drops) and the cut-off point is 200ng/ml. Urine tests can be traced up to 7-10 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Inha University Hospital, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: Undecided